CLINICAL TRIAL: NCT01872845
Title: A Trial Comparing the Effect of Pravastatin and Rosuvastatin on Atherosclerosis Progression Measured by Carotid Intima Media Thickness in Patients With Coronary Artery Disease After Biolimus Eluting Stent (Nobori®) Implantation: CPR IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0206
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Occlusive Disease
Keywords: Statin; CIMT; BES
MeSH Terms: interventions — Pravastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Active Comparator): All study subjects will be received percutaneous coronary intervention (PCI) with Biolimus-eluting stent as index procedure at the time of enrollment After index procedure, patients will be randomly assigned to receive pravastatin 40mg or rosuvastatin 20mg in a 1:1 ratio. a> Test group: Pravastatin 40mg PO daily for 1year from the day of BES implantation b> Control group: Rosuvastatin 20mg PO daily for 1year from the day of BES implantation
  Interventions: Drug: Rosuvastatin
- Pravastatin (Experimental): All study subjects will be received percutaneous coronary intervention (PCI) with Biolimus-eluting stent as index procedure at the time of enrollment After index procedure, patients will be randomly assigned to receive pravastatin 40mg or rosuvastatin 20mg in a 1:1 ratio. a> Test group: Pravastatin 40mg PO daily for 1year from the day of BES implantation b> Control group: Rosuvastatin 20mg PO daily for 1year from the day of BES implantation
  Interventions: Drug: Pravastatin 40mg

INTERVENTIONS:
Drug: Pravastatin 40mg — Pravastatin 40mg PO daily for 1year from the day of BES implantation
  Arms: Pravastatin
Drug: Rosuvastatin — Rosuvastatin 20mg PO daily for 1year from the day of BES implantation
  Arms: Rosuvastatin

SUMMARY:
Current consensus papers recommend statin medication to reduce Low density lipoprotein (LDL) cholesterol level less than 100mg/dL (optional 70mg/dL) in patients with coronary artery disease. However, there is lack of solid evidence whether a specific kind of statin have the superiority against other statins in clinical outcomes. Furthermore, recent data have showed that several kinds of statin could have an adverse effect on glucose metabolism and increase the risk of development of diabetes. Carotid Intimamedia thickness (CIMT) is a surrogate marker of atherosclerosis to predict long term cardiovascular outcomes in not only general population but also patients with established coronary artery disease. Consequently, we will evaluate the efficacy of high dose of pravastatin on CIMT, comparing with moderate dose of rosuvastatin in patients with established coronary artery disease. Additionally, we will assess the clinical outcomes of pravastatin after percutaneous coronary intervention as well as adverse outcomes including insulin resistance and new onset diabetes compared with rosuvastatin. Our main hypothesis is that pravastatin 40mg would be non-inferior to rosuvastatin 20mg regarding CIMT at 1 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 20 years old
* Patients with coronary artery disease who are candidate for coronary revascularization with DES implantation.
* Significant coronary de novo lesion (stenosis > 70% by quantitative angiographic analysis)
* Patients eligible for statin treatment (initial LDL cholesterol >70mg/dL or patients taking lipid-lowering agent)

Exclusion Criteria:

* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Change of carotid intima media thickness 1 year after pravastatin or rosuvastatin treatment | 1 year after drug-eluting stent implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea